CLINICAL TRIAL: NCT00026286
Title: A Phase III Prospective, Randomized, Double-Blind Clinical Trial of Hormone Replacement Therapy In Postmenopausal Women With A History Of Node-Negative Or Ductal Carcinoma In Situ Who Are Receiving Adjuvant Tamoxifen
Brief Title: Hormone Replacement Therapy for Hot Flashes and/or Vaginal Symptoms in Postmenopausal Women Receiving Tamoxifen for Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000069015; E-2193; NCI-P01-0194
Record Dates: First submitted 2001-11-09; First posted 2003-09-17 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer; Hot Flashes; Menopausal Symptoms
Keywords: stage I breast cancer; stage II breast cancer; breast cancer in situ; ductal breast carcinoma; hot flashes; menopausal symptoms
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes; Breast Carcinoma In Situ; Carcinoma, Ductal, Breast | interventions — Estrogens, Conjugated (USP); Medroxyprogesterone

INTERVENTIONS:
Drug: conjugated estrogens
Drug: medroxyprogesterone

SUMMARY:
RATIONALE: Hormone replacement therapy may be effective in managing the hot flashes and/or vaginal symptoms in postmenopausal women who are receiving tamoxifen for breast cancer.

PURPOSE: Randomized phase III trial to determine the effectiveness of hormone replacement therapy in managing hot flashes and/or vaginal symptoms in postmenopausal women who are receiving tamoxifen for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of hormone replacement therapy in managing hot flashes and menopausal vaginal symptoms in postmenopausal women with a history of node-negative invasive carcinoma or ductal carcinoma in situ of the breast who are receiving adjuvant tamoxifen.
* Determine the effect of this regimen on blood coagulation and lipid profiles in these patients.
* Determine the quality of life of patients treated with this regimen.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to prior hysterectomy (yes vs no), symptom complex (vasomotor vs vaginal vs both), duration of hot flashes (less than 1 year or no hot flashes vs 1 year or more), and average daily number of hot flashes (less than 10 or none vs 10 or more). Patients are randomized to one of two treatment arms.

* Arm I: Patients who have not undergone prior hysterectomy receive oral medroxyprogesterone once daily for 6 months. If, after 1 month, symptoms do not resolve, patients receive oral conjugated estrogens once daily in addition to medroxyprogesterone for 5 months. Patients who have undergone prior hysterectomy receive oral conjugated estrogens once daily for 6 months.
* Arm II: Patients receive oral placebo once daily for 6 months. Quality of life is assessed at baseline and months 1, 2, 3, and 6.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 120 patients (60 per treatment arm) will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed node-negative invasive carcinoma or ductal carcinoma in situ of the breast
* No contralateral breast cancer
* No recurrent or metastatic disease
* Completion of active non-hormonal therapy for breast cancer
* Receiving tamoxifen (20 mg/day) for at least 3 months prior to study and plan to continue drug while on study
* Hot flashes severe enough to seek medical intervention (at least 7-8 moderate to severe hot flashes per day or 60 per week at baseline) AND/OR
* Vaginal symptoms, including dyspareunia, vaginal dryness, irritation, or thinning due to estrogen deficiency
* If uterus present, no prior histologically confirmed adenomatous or atypical endometrial hyperplasia or endometrial carcinoma AND no concurrent endometrial cancer confirmed by pelvic exam within the past year
* No active endometriosis
* No unexplained vaginal bleeding
* Hormone receptor status:

  * Estrogen and progesterone receptor status known for patients with invasive breast cancer

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Postmenopausal
* No menstrual period for more than 12 months OR prior bilateral oophorectomy
* Must be over 55 years of age OR have documented follicle-stimulating hormone levels in postmenopausal range if one or both ovaries remain after prior hysterectomy

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No prior superficial or deep venous or arterial thrombosis
* No serious venous stasis disease

Pulmonary:

* No pulmonary embolus

Other:

* Must be able to read and speak English
* No lower extremity trauma, swelling, or tenderness within the past 4 weeks
* No active gallbladder disease
* No migraine headaches
* No other prior malignancy unless curatively treated with no evidence of recurrence
* No concurrent seizure disorder requiring anti-seizure medication

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* See Disease Characteristics
* No other concurrent estrogen or hormone replacement therapy
* No concurrent clonidine, bellergal, progestational agent, or methyldopa for hot flashes
* No concurrent topical vaginal estrogen cream (e.g., Estring or Vagifem) for patients with vaginal symptoms only

Radiotherapy:

* Not specified

Surgery:

* At least 4 weeks since prior surgery

Other:

* At least 12 months since prior treatment for congestive heart failure
* Concurrent selective serotonin reuptake inhibitors (SSRI) or antidepressants with SSRI activity allowed if begun at least 3 months prior to study and continue during study

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-11-28 (Actual); Primary Completion 2002-08 (Actual); Study Completion 2007-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melody A. Cobleigh, MD, Study Chair — Rush University Medical Center
Locations (24):
- United States (24):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Veterans Affairs Medical Center - Tennessee Valley Healthcare System - Nashville Campus, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin